

F-INV001 V: 03

Date of Writing/Update: Octuber 2024

Project version: 1.0

Clinical Effectiveness, Adherence, Clinical and Paraclinical Outcomes Associated with Tenofovir Alafenamide/Emtricitabine/Bictegravir (TAF/FTC/BIC) in Patients Diagnosed with Human Immunodeficiency Virus (HIV) in Colombia: A Real-Life Study

### **Research Question**

What are the clinical effectiveness, adherence, and clinical and paraclinical outcomes associated with Tenofovir Alafenamide/Emtricitabine/Bictegravir (TAF/FTC/BIC) in patients diagnosed with HIV in a Colombian EPS?

- P (Population): Patients aged 18 years and older diagnosed with HIV.
- I (Intervention): Treatment with TAF/FTC/BIC.
- C (Comparison): N/A.
- (Outcomes): Clinical effectiveness, adherence, and clinical and paraclinical outcomes.

### **Summary**

HIV remains one of the most serious global pandemics, affecting 38 million people, with the highest prevalence in sub-Saharan Africa. Stigma and discrimination continue to hinder diagnosis and treatment, impacting marginalized populations most significantly. In Latin America, prevalence remains stable at approximately 0.4%, though Colombia faces unique challenges, with an epidemic concentrated among men who have sex with men. Recently published high-cost data from Colombia indicate that there are currently 165,405 people living with HIV (PLHIV), with 14,670 new cases reported in 2023. Social and economic factors, along with Venezuelan migration, complicate access to treatment in Colombia.

F-INV001 V: 03

Advances in ART have been made with the use of integrase inhibitors such as TAF/FTC/BIC, which has demonstrated effectiveness across various populations. However, real-world studies specific to Colombia are lacking. In this study, we aim to evaluate adherence, effectiveness, and clinical outcomes of TAF/FTC/BIC treatment in a cohort of 169 patients within a larger group of 15,300 HIV patients under the EPS SURA program, generating evidence that is relevant to the Colombian context.

#### **Problem Statement and Relevance**

HIV remains one of the most significant global pandemics, with approximately 38 million people living with HIV worldwide, according to medical literature. The prevalence is particularly high in sub-Saharan Africa, which accounts for 70% of infections (1-3). Additionally, HIV is a leading cause of disability-adjusted life years (DALYs), ranking as the fifth leading cause globally in 2010 (4).

Stigma and discrimination remain major barriers to the diagnosis and treatment of HIV, disproportionately affecting marginalized populations such as sex workers, people who inject drugs, men who have sex with men, and transgender individuals (5). Despite advances in treatment, HIV remains a chronic condition that requires lifelong drug therapy to suppress viral load and prevent transmission (6).

In Latin America, HIV infection is recognized as a public health issue with unique epidemiological characteristics and challenges that vary across the region. HIV prevalence is relatively stable in Latin America, averaging 0.4% in the general population, though significant differences exist both between and within countries. Brazil, Mexico, and Colombia have the highest number of cases (7,8). In the Caribbean, for example, prevalence among adults exceeds 1% in several countries, where a decrease in new infections has also been observed (8).

F-INV001 V: 03

HIV infection in Colombia poses a significant public health challenge, as the country has the fourth highest incidence rate of HIV/AIDS in Latin America, which has been rising since the 1980s (9). The epidemic is concentrated within key populations, such as men who have sex with men, who bear a high HIV burden in the country's major cities, with prevalence ranging from 6% to 24% (10). In 2023, 14,603 new cases were reported, marking a 13.5% increase compared to 2022. Of these cases, 34% were diagnosed at the AIDS stage. This trend of rising incidence and late diagnoses has been observed since the COVID-19 pandemic, likely due to delayed healthcare access. In 2023, new diagnoses in men accounted for 83% of cases compared to women.

HIV transmission in Colombia is influenced by social and economic factors, including social inequalities and sex tourism, particularly in cities like Cartagena (11). Co-infection with the hepatitis C virus is also becoming a growing issue among people living with HIV. Of the 1,058 new cases of hepatitis C reported in Colombia in 2023, 69.47% were co-infected with HIV (12). Additionally, hepatitis C is emerging as a significant problem among people who inject drugs (13). While access to antiretroviral therapy (ART) has improved, significant barriers to early diagnosis and timely treatment remain, exacerbated by social stigma, limited access to healthcare, and the impact of large-scale migration from Venezuela. This migration has placed added pressure on the Colombian healthcare system and disrupted the continuity of care for migrants living with HIV (14,15).

Current recommendations for the initiation of antiretroviral therapy (ART) include the use of an integrase strand transfer inhibitor (INSTI), such as bictegravir or dolutegravir, in combination with a nucleoside reverse transcriptase inhibitor (NRTI). These options have proven to be effective, with a high genetic barrier and potent activity in infected patients (16,17). Bictegravir/Emtricitabine/Tenofovir Alafenamide (TAF/FTC/BIC) is a single-tablet combination therapy developed for the treatment of HIV. Its mechanism of action combines the INSTI bictegravir with the NRTIs emtricitabine and tenofovir alafenamide,



F-INV001 V: 03

demonstrating efficacy in both treatment-naïve patients (those without prior exposure to ART) and patients previously exposed to ART (18).

As of January 2024, EPS SURA manages a cohort of approximately 15,300 HIV patients. The control, evaluation, and follow-up of these patients are primarily conducted by specialized healthcare institutions (IPS), with a smaller proportion monitored by affiliated IPS providers. Program indicators include treatment abandonment rates, virological success rates, virological success with ART in the last 3 months, HIV viral load, and CD4 T-lymphocyte levels in the past 6 months for patients with HIV. To assess patient adherence, regular weekly evaluations are conducted, which include laboratory monitoring and attendance at medical appointments. In cases of non-compliance, a strict follow-up plan is established by a designated physician and a pharmaceutical chemist to verify medication intake and evaluate risk factors associated with non-adherence on an individual basis. From 2020 to 2023, 169 patients within the HIV program were prescribed TAF/FTC/BIC treatment.

To date, few studies have been conducted in real-life conditions (19-22) to evaluate the effectiveness, safety, and clinical outcomes of TAF/FTC/BIC initiation, especially in patients at later stages of HIV, in everyday contexts. These outcomes are influenced by factors such as timely access to healthcare, follow-up, and proper adherence. No real-life studies have been conducted in Colombia, despite integrase inhibitors being the first-line treatment in the country and widely available as part of the mandatory health plan. Therefore, it is essential to evaluate the effectiveness, adherence, and clinical outcomes within our cohort. Generating our own data will allow us to create evidence with significant population impact.

### Theoretical framework

Human Immunodeficiency Virus (HIV) is a retrovirus from the Retroviridae family,



F-INV001 V: 03

specifically an enveloped positive-stranded RNA virus (5). There are two main types: HIV-1, the most common worldwide, and HIV-2, which is more prevalent in West Africa (23). The virus is transmitted through bodily fluids such as blood, semen, vaginal secretions, and breast milk. Once inside the body, HIV primarily targets CD4+ T lymphocytes of the immune system, binding to CD4 receptors and one of the chemokine co-receptors, CCR5 or CXCR4, to enter the host cell (6). This process of viral entry and replication leads to the progressive destruction of CD4+ T lymphocytes, resulting in severe immunodeficiency if not treated promptly (6,24).

The molecular structure of HIV includes several key proteins. The virus is enveloped by a lipid membrane containing envelope glycoproteins (Env), specifically gp120 and gp41, which form a functional trimer. These glycoproteins are crucial for binding and fusion with host cells. Gp120 binds to the CD4 receptor on the surface of T lymphocytes, causing conformational changes that allow it to interact with the CCR5 or CXCR4 co-receptors, facilitating viral entry (25-27).

Its genome is RNA-based and encodes 15 distinct proteins, including structural Gag proteins (MA, CA, NC, p6), Pol enzymes (protease, reverse transcriptase, integrase), and accessory and regulatory proteins such as Tat, Rev, Nef, Vif, Vpr, and Vpu (28). These proteins play critical roles in the viral life cycle, from entry to replication and assembly (26,28). While HIV-1 and HIV-2 share structural similarities, they also exhibit significant differences in their envelope glycoproteins, which influence their pathogenicity and immune response. For example, HIV-2 has lower pathogenicity and a greater capacity to induce neutralizing antibodies (29,30). These structural and functional characteristics are crucial for understanding the mechanism of infection and for developing therapeutic and prevention strategies, such as vaccines (25,26).

### Pathophysiology of HIV

The pathophysiology of HIV involves a series of complex mechanisms that result in

F-INV001 V: 03

progressive immunosuppression (31-33). The process begins with the binding of the HIV envelope glycoprotein to the CD4 receptor on the surface of CD4+ T lymphocytes and other cells, such as macrophages (31). This facilitates virus entry and replication within host cells. During primary infection, acute viremia occurs with extensive viral shedding, and the virus is sequestered in the germinal centers of lymphoid tissues (34). There is massive destruction of memory CD4+ T lymphocytes early in the infection, although this does not initially lead to overt immunodeficiency. However, over time, the regeneration of these cells proves insufficient, resulting in the failure of immune homeostasis and progression to AIDS (Acquired Immunodeficiency Syndrome) (32,33).

In addition, chronic immune activation and immune dysfunction contribute significantly to the pathogenesis of the virus. Inappropriate activation of the immune system and the elevated secretion of proinflammatory cytokines regulate HIV expression in tissues (34). Infection of progenitor cells in the bone marrow and thymus also contributes to the impaired regeneration of immunocompetent cells (34). Furthermore, HIV causes direct damage to various tissues, such as the gut, brain, and lungs, through infection and activation of mononuclear cells (24). Systemic immune response activation and the destruction of lymphoid follicle integrity are hallmark features of pathogenic infection (35).

### Clinical Manifestations of HIV

The clinical manifestations of HIV are varied and affect multiple systems due to the progressive immunosuppression and chronic immune activation that characterize the infection. HIV can be divided into several clinical phases, each with distinct characteristics:

- Acute infection: This phase occurs within the first few weeks after exposure to the virus. Symptoms may include fever, adenopathy, pharyngitis, rash, myalgias, and arthralgias. This phase resembles an acute viral syndrome and is often underdiagnosed (36,37).
- 2. Chronic asymptomatic phase: Many patients enter a clinical latency phase that can last for several years. During this time, the virus continues to replicate and destroy



F-INV001 V: 03

CD4+ T cells, but patients may remain asymptomatic (36,37).

- 3. Advanced Immunosuppression and AIDS: As the infection progresses and CD4+ T-lymphocyte counts decline, patients become increasingly susceptible to opportunistic infections and neoplasms. Common opportunistic infections include Pneumocystis jirovecii pneumonia, esophageal candidiasis, cytomegalovirus disease, cerebral toxoplasmosis, and pulmonary or disseminated tuberculosis, among others. The prevalence of these infections varies depending on the degree of immunosuppression and the geographical region. Some neoplasms associated with HIV include Kaposi's sarcoma, non-Hodgkin's lymphoma, and invasive cervical cancer (24,36,37).
- 4. Non-Infectious Manifestations: HIV is also linked to a range of non-infectious complications due to chronic immune activation and systemic inflammation. These include cardiovascular, hepatic, renal, bone, and neurological diseases. Cardiovascular disease in HIV patients may manifest as coronary artery disease, dilated cardiomyopathy, pulmonary hypertension, and endothelial dysfunction. Liver complications may involve virus-associated viral hepatitis and drug-induced hepatotoxicity, while renal dysfunction can present as HIV-associated nephropathy (37-39).
- 5. Hematological Manifestations: These are common and may include anemia, leukopenia, and thrombocytopenia. These conditions may result from the direct infection of hematopoietic progenitor cells, bone marrow dysfunction, and activation of the reticuloendothelial system (40).
- 6. Immune Reconstitution Inflammatory Syndrome (IRIS): In patients initiating ART, a paradoxical exacerbation of underlying infections may occur due to partial recovery of the immune system. IRIS can complicate clinical management and requires careful monitoring (24,41). In some cases, ART initiation should be postponed for a few weeks, especially when diagnosing opportunistic infections such as cytomegalovirus disease or meningeal cryptococcosis, to avoid exacerbation or worsening of symptoms, which can lead to considerable morbidity



F-INV001 V: 03

and mortality.

## Diagnosis of HIV

HIV diagnosis is performed using a combination of tests that detect viral RNA, p24 antigen, and HIV-specific antibodies. This approach allows for the identification of both acute and chronic infections:

- HIV RNA: Detection of viral RNA is possible approximately 10-12 days after exposure to the virus, making this test particularly useful in the acute phase of infection, when antibodies are not yet detectable (23).
- 2. p24 Antigen: The p24 antigen appears in serum or plasma about 15-17 days after exposure. Detection of p24 antigen is a key feature of fourth- and fifth-generation tests, which allow for the identification of infection before antibodies develop (5,23).
- 3. Specific Antibodies: HIV antibodies (IgM and IgG) are detectable in serum or plasma approximately 21 days after exposure. Today, fourth-generation tests combine antibody detection with p24 antigen detection, improving sensitivity and enabling earlier detection of infection (5,42,43).

The diagnostic algorithm recommended by the CDC in the United States begins with a laboratory antigen/antibody (Ag/Ab) combination test. If this test is reactive, it is followed by an antibody differentiation test to distinguish between HIV-1 and HIV-2. If the differentiation test is negative or indeterminate, a nucleic acid amplification test is conducted to confirm acute infection (43,44). In Colombia, there is also a diagnostic algorithm that begins with a first rapid test (ELISA, chemiluminescence, or molecular test). If the first test is reactive, a second test should be performed to confirm the diagnosis. In cases of discordance, a molecular test for RNA detection or the Western Blot technique can be used (45).

### **HIV Treatment**

It is critical that HIV treatment be initiated as early as possible (45). There is substantial

F-INV001 V: 03

medical evidence that early initiation of ART prevents complications related to immunosuppression and reduces mortality. Treatment requires lifelong ART, which has transformed a fatal disease into a manageable chronic condition. Modern ART consists of combinations of at least three drugs from two or more different classes, providing long-lasting virologic suppression and improving clinical outcomes (46,47). Regimen selection is based on factors such as virologic efficacy, adverse effect profiles, pill burden, dosing frequency, drug-drug interactions, resistance test results, comorbidities, and cost (46).

In low- and middle-income countries, access to this therapy remains uneven due to economic constraints, inadequate health infrastructure, and social stigmatization (48,49). Despite these challenges, global efforts have enabled millions of people in these regions to access life-saving treatment (49). However, significant barriers to achieving universal coverage remain, including the need for improved early detection and timely initiation of treatment (50).

Recent innovations in ART include the development of drugs with improved safety and resistance profiles, as well as combination therapies that enhance adherence, such as single-tablet regimens and long-acting ARVs (46,47). These advances are particularly promising for improving adherence and reducing treatment burdens in low- and middle-income countries (50). Additionally, research into curative therapies, such as latency reversal agents and gene therapy, is ongoing, although their implementation faces challenges due to differences in host genetics and viral subtypes (48,51).

Bictegravir is a second-generation integrase strand transfer inhibitor (INSTI) used in HIV treatment. It is a key component of BikARVTy®, a fixed-dose regimen combining bictegravir, emtricitabine, and tenofovir alafenamide in a single daily tablet (52,53). This drug is notable for its high genetic barrier to resistance, meaning the virus is less likely to develop resistance to it compared to other INSTIs such as raltegravir and elvitegravir (54,55). It also has a limited drug-drug interaction profile, making it suitable for use in



F-INV001 V: 03

combination with other antiretrovirals (52,56).

In phase 3 clinical trials, the bictegravir/emtricitabine/tenofovir alafenamide regimen has been shown to be non-inferior to dolutegravir-based regimens in both treatment-naïve and treatment-experienced patients, achieving effective virologic suppression without the emergence of resistance (53,57,58). Additionally, it is well tolerated and does not require prior HLA-B\*5701 testing, which facilitates its rapid initiation in HIV treatment (53,57).

The most common adverse effects reported in clinical trials include diarrhea, nausea, and headache, with an incidence of at least 5% in treated subjects (59). Other less frequent adverse effects (≥2%) include fatigue, abnormal dreams, dizziness, insomnia, and abdominal distension (59). Regarding laboratory abnormalities, increases in serum creatinine, which stabilized throughout treatment, and increases in total bilirubin, mainly grade 1 and 2, were observed. Most adverse events were grade 1, and discontinuations due to adverse events were uncommon (59). Psychiatric events, such as suicidal ideation and depression, have also been reported, particularly in subjects with a history of psychiatric conditions. In subjects with end-stage renal disease, serious adverse events such as pneumonia and fluid overload were observed (59).

### **Objectives**

**General Objective:** To estimate the clinical effectiveness and safety of HIV-positive patients on TAF/FTC/BIC treatment within an EPS in Colombia.

## **Specific Objectives:**

- To characterize the sociodemographic and clinical profile of patients with HIV who initiate antiretroviral therapy with TAF/FTC/BIC.
- To identify the proportion of patients who have been on different pretreatment regimens before initiating TAF/FTC/BIC therapy.
- To assess the proportion of patients achieving virologic suppression at weeks 24



F-INV001 V: 03

and 48 following the initiation of TAF/FTC/BIC therapy.

- To determine the proportion of patients with effective access to TAF/FTC/BIC therapy.
- To describe the impact of TAF/FTC/BIC treatment on CD4+ T-lymphocyte count, renal function, and lipid profile at weeks 24 and 48 after starting therapy.
- To determine the proportion of patients with a rapid onset of TAF/FTC/BIC therapy.
- To characterize the proportion of treatment-related adverse events at weeks 24 and 48 after initiating TAF/FTC/BIC therapy.
- To identify the proportion of patients meeting the criteria for adherence to TAF/FTC/BIC therapy.

### Methodology

## Study Design

This is an observational, retrospective cohort study that will include adult patients who received treatment with TAF/FTC/BIC between January 2020 and December 2023. The study will include both treatment-naïve patients and those who have been previously exposed to other treatments. The index date will correspond to the initiation date of the drug, at which point baseline demographic and clinical characteristics will be recorded.

### Data Collection Plan/Source Documents

SURA is one of Colombia's leading insurers and has an integrated network of care centers. The clinical and administrative records of all its affiliates are stored in a centralized digital information system, which includes both structured and unstructured data. Data collection will be conducted through a retrospective review of electronic medical records, using a pre-designed Excel database (with an institutional Office license). This database will include the variables defined in the project. The study will utilize secondary data collected from the electronic records generated for each patient during the provision of health services. The conversion of unstructured data into structured



F-INV001 V: 03

data during the execution of the protocol will be done solely through automated/algorithmic methods on a computer. To ensure consistency and standardization, the template will be parameterized with predefined answers or options for each variable. These will be defined based on medical experience, the availability of information, and in accordance with the protocol's guidelines.

All data will undergo a cleaning process, evaluating four key aspects: consistency, completeness, validity, and uniformity. Consistency is checked to ensure that the data are coherent and that harmonized codes and labels are used. Completeness ensures that the data are fully filled out and ready for use. Validity verifies that the data meet the required standards and fall within the established range. Uniformity ensures that the data are not duplicated and cannot be confused with other entries.

Subsequently, all relevant information will be extracted, creating a copy of the original record, which will be sent to the requester in tabular format (Microsoft Excel). The principal investigator or their delegate will import the Excel file into RStudio and Jamovi. Unstructured data will be obtained through a manual search of the patients' medical records, ensuring that the information is accurate, authentic, attributable, complete, consistent, legible, timely, and durable. These will be manually recorded in a flat file (Microsoft Access) and subsequently transferred to RStudio and Jamovi for analysis.

The following ICD-10 codes are considered key data for searching patient medical records:

- B200: HIV disease resulting in mycobacterial infection.
- B201: HIV disease resulting in other bacterial infections.
- B202: HIV disease resulting in cytomegalovirus disease.
- B203: HIV disease resulting in other viral infections.
- B204: HIV disease resulting in candidiasis.
- B205: HIV disease resulting in other mycoses.



F-INV001 V: 03

- B206: HIV disease resulting in *Pneumocystis carinii* pneumonia.
- B207: HIV disease resulting in multiple infections.
- B208: HIV disease resulting in other infectious or parasitic diseases.
- B209: HIV disease resulting in unspecified infectious or parasitic disease.
- B210: HIV disease resulting in Kaposi's sarcoma.
- B211: HIV disease resulting in Burkitt's lymphoma.
- B212: HIV disease resulting in other types of non-Hodgkin's lymphoma.
- B213: HIV disease resulting in other malignant tumors of lymphoid, hematopoietic, and related tissues.
- B217: HIV disease resulting in multiple malignant tumors.
- B218: HIV disease resulting in other malignant tumors.
- B219: HIV disease resulting in unspecified malignant tumors.
- B220: HIV disease resulting in encephalopathy.
- B221: HIV disease resulting in lymphoid interstitial pneumonitis.
- B222: HIV disease resulting in cachectic syndrome.
- B227: HIV disease resulting in multiple illnesses classified elsewhere.
- B230: Acute HIV infection syndrome.
- B231: HIV disease resulting in generalized lymphadenopathy (persistent).
- B232: HIV disease resulting in immunologic and hematologic abnormalities, not elsewhere classified.
- B238: HIV disease resulting in other specified conditions.
- B24X: Human immunodeficiency virus (HIV) disease, not otherwise specified.
- F024: Dementia in human immunodeficiency virus (HIV) disease (B22.0†).
- Z21X: Asymptomatic human immunodeficiency virus (HIV) infection status.

All information on the variables of interest will be extracted from the clinical records. The process of data collection and form completion will be carried out by personnel from the Clinical Research Unit, following training to ensure standardized data capture. Quality



F-INV001 V: 03

control of the data will be performed, including the review of codes, missing data, and any incorrect or improperly transcribed characters, according to the variable, by the researchers before the dataset is purified for analysis.

### Study Population

All patients who meet the defined selection criteria within the established time frame for the search will be included:

- Inclusion Criteria:
  - Male or female patients aged 18 years or older.
  - Individuals with a confirmed HIV diagnosis.
  - o Individuals enrolled in EPS SURA during the study period.
  - o Patients receiving treatment with the TAF/FTC/BIC regimen.
- Exclusion Criteria:
  - Patients with a concurrent diagnosis of tuberculosis.
  - Pregnant patients during the study period.
  - Patients with virologic failure.
  - Patients who started treatment with TAF/FTC/BIC but changed providers or discontinued treatment before completing six months of therapy.

#### Variables

| Variable Name | Definition | Nature | Measuring Level |
|---|---|---|---|
| Primary diagnosis of HIV | Patient with primary ICD-10 diagnosis of: B200, B201, B202, B203, B204, B205, B206, B207, B208, B209, B210, B211, B212, B213, B217, B218, B219, B220, B221, B222, B227, B230, B231, B232, B238, B24X, F024 or Z21X | Qualitative | Text |
| Diagnosis date | Date of first confirmed repeat HIV diagnosis recorded in the medical record | Quantitative, continuous | dd/mm/yyyy |
| Date of birth | pirth Patient's date of birth Quantitative continuous | | dd/mm/yyyy |
| Sex | Sex defined by patient's medical history Qualitative | | 0: Female; 1:<br>Male. |
| Race | Race defined by patient's medical history | Qualitative | Texto |



| Type of insurance | Insurance from the health system to whom the patient is covered. Qualitative | | 0: Public<br>1: Private |
|---|---|---|---|
| Residence department | Department of Colombia where the patient lives | Qualitative | Text |
| AHT | Patient with hypertension marked in electronic medical record | Qualitative | 0: No<br>1: Yes |
| Diabetes Mellitus | Patient with diabetes marked in electronic medical record | Qualitative | 0: No<br>1: Yes |
| Chronic kidney disease | Patient with chronic kidney disease marked in electronic medical record | Qualitative | 0: No<br>1: Yes |
| Hepatitis B co-infection | Patient with repeated confirmed ICD-10 diagnosis of B181 Chronic type B viral hepatitis, no delta agent from the date of HIV diagnosis to the end of follow-up. | Qualitative | 0: No<br>1: Yes |
| Hepatitis C co-infection | Patient with repeated confirmed ICD-10 diagnosis of B182 Chronic viral hepatitis type C from the date of HIV diagnosis to the end of follow-up. | epeated confirmed ICD-10 32 Chronic viral hepatitis type of HIV diagnosis to the end Qualitative | |
| Major depressive disorder | Patient with confirmed ICD-10 repeat diagnoses: F320, F321, F322, F323, F328, F329, F330, F331, F332, F333, F334, F338, F339, F340, F341, F348, F349, F380, F381, F388 or F39X from the date of HIV diagnosis to the end of follow-up | | 0: No<br>1: Yes |
| Start date TAF/FTC/BIC | Medication start date TAF/FTC/BIC | Quantitative, continuous | dd/mm/yyyy |
| End date TAF/FTC/BIC | Medication end date TAF/FTC/BIC | Quantitative, continuous | dd/mm/yyyy |
| NAIVE for TAF/FTC/BIC | Patient whose first HIV treatment is TAF/FTC/BIC | Qualitative | 0: No<br>1: Yes |
| ARVT scheme prior to TAF/FTC/BIC | Name of ARVT scheme immediately preceding TAF/FTC/BIC used for HIV treatment | Qualitative | Text |
| HIV viral load at baseline | The patient has HIV viral load results at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy. | Qualitative | 0: No<br>1: Yes |
| BHIV viral load at baseline value | HIV viral load value at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| HIV viral load at week 24 | The patient has HIV viral load results at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | Qualitative | 0: No<br>1: Yes |
| HIV viral load value at week 24 | HIV viral load value at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| HIV viral load at week 48 | The patient has HIV viral load results at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | Qualitative | 0: No<br>1: Yes |
| HIV viral load value at week 48 | HIV viral load value at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| CD4 Lymphocyte count at baseline | The patient has CD4 Lymphocyte count results at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy. | Qualitative | 0: No<br>1: Yes |
| CD4 Lymphocyte count at baseline value | count at CD4 Lymphocyte count value at baseline (+ Cu | | 1, 1.5, 1.8, 2, n |



| CD4 Lymphocyte count at week 24 | The patient has CD4 Lymphocyte count results at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | | 0: No<br>1: Yes |
|---|---|---|---|
| CD4 Lymphocyte count value at week 24 | CD4 Lymphocyte count value at week 24 (+ or - 2 weeks) of therapy with TAF/FTC/BIC | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| CD4 Lymphocyte count at week 48 | The patient has CD4 Lymphocyte count results at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | Qualitative | 0: No<br>1: Yes |
| CD4 Lymphocyte count value at week 48 | CD4 Lymphocyte count value at week 48 (+ or - 2 weeks) of therapy with TAF/FTC/BIC | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| HDL at baseline | The patient has high-density lipoprotein results at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy | Qualitative | 0: No<br>1: Yes |
| HDL value at baseline | High-density lipoprotein value at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| HDL at week 24 | The patient has high-density lipoprotein results at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | | 0: No<br>1: Yes |
| HDL value at week 24 | High-density lipoprotein value at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| HDL at week 48 | The patient has high-density lipoprotein results at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | 0: No<br>1: Yes | |
| HDL value at week 48 | High-density lipoprotein value at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy continuous | | 1, 1.5, 1.8, 2, n |
| LDL at baseline | The patient has low-density lipoprotein at baseline results at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy. Qualitative | | 0: No<br>1: Yes |
| LDL value at baseline | Low-density lipoprotein value at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| LDL at week 24 | The patient has low-density lipoprotein HDL results at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | Qualitative | 0: No<br>1: Yes |
| LDL value at week 24 | Low-density lipoprotein HDL value at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| LDL at week 48 | The patient has low-density lipoprotein results at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | | 0: No<br>1: Yes |
| LDL value at week 48 | Low-density lipoprotein value at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| AST at baseline | The patient has aspartate aminotransferase results at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy. | Qualitative | 0: No<br>1: Yes |
| AST at baseline value | Aspartate aminotransferase value at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| AST at week 24 | The patient has aspartate aminotransferase results at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | | 0: No<br>1: Yes |
| AST value at week 24 | Aspartate aminotransferase value at week 24 | | 1, 1.5, 1.8, 2, n |



| AST at week 48 | The patient has aspartate aminotransferase results at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | 0: No<br>1: Yes | |
|---|---|---|---|
| AST value at week 48 | Aspartate aminotransferase value at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| ALT at baseline | The patient has alanine aminotransferase results at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy. | Qualitative | 0: No<br>1: Yes |
| ALT value at baseline | Alanine aminotransferase value at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| ALT week at 24 | The patient has alanine aminotransferase results at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy. | Qualitative | 0: No<br>1: Yes |
| ALT value week at 24 | Alanine aminotransferase level at week 24 (+ or – 2 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| ALT week at 48 | The patient has alanine aminotransferase results at week 48 (+ or - 2 weeks) of therapy with TAF/FTC/BIC. | | 0: No<br>1: Yes |
| ALT value at week 48 | Alanine aminotransferase value at week 48 (+ or - 2 weeks) of therapy with TAF/FTC/BIC. | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| Total bilirubin at baseline | The patient has total bilirubin results at baseline (+ or - 4 weeks) of therapy with Cualitative TAF/FTC/BIC. | | |
| Total bilirubin value at baseline | Total bilirubin value at baseline (+ or - 4 weeks) of therapy with TAF/FTC/BIC. | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| Total bilirubin at week 24 | The patient has total bilirubin results at week 24 (+ or - 2 weeks) of therapy with TAF/FTC/BIC. | Qualitative | 0: No<br>1: Yes |
| Total bilirubin value at at week 24 | Total bilirubin value at week 24 (+ or - 2 weeks) of therapy with TAF/FTC/BIC. | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| Total bilirubin at week 48 | The patient has total bilirubin results at week 48 (+ or – 2 weeks) of TAF/FTC/BIC therapy | Qualitative | 0: No<br>1: Yes |
| Total bilirubin value at week 48 | Total bilirubin value at week 48 (+ or – 2 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| Serum creatinine at baseline | The patient has baseline serum creatinine results (+ or – 4 weeks) of TAF/FTC/BIC therapy | Qualitative | 0: No<br>1: Yes |
| Serum creatinine value at baseline | Baseline serum creatinine value (+ or – 4 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| Serum creatinine at week 24 | - Week 24 (+ or - 2 weeks) of TAF/FTC/BIC T QUAINATIVE | | 0: No<br>1: Yes |
| Serum creatinine value at week 24 | Serum creatinine value at week 24 (+ or – 2 Quantii weeks) of TAF/FTC/BIC therapy contin | | 1, 1.5, 1.8, 2, n |
| Serum creatinine at week 48 | The patient has serum creatinine results at week 48 (+ or – 2 weeks) of TAF/FTC/BIC Qualitative therapy | | 0: No<br>1: Yes |
| Serum creatinine value at week 48 | reatinine value at Serum creatinine value at week 48 (+ or – 2 | | 1, 1.5, 1.8, 2, n |

F-INV001 V: 03

| Glomerular filtration rate at baseline | The patient has the estimated glomerular filtration rate (eGFR) by CKD-EPI at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy | Qualitative | 0: No<br>1: Yes |
|---|---|---|---|
| Value of glomerular filtration rate at baseline | Value of estimated glomerular filtration rate (eGFR) calculated by CKD-EPI at baseline (+ or - 4 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| Glomerular filtration rate at week 24 | The patient has an estimated glomerular filtration rate (eGFR) calculated by CKD-EPI at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy | Qualitative | 0: No<br>1: Yes |
| Glomerular filtration rate value at week 24 | Value of estimated glomerular filtration rate (eGFR) calculated by CKD-EPI at week 24 (+ or - 2 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| Glomerular filtration rate at week 48 | The patient has the estimated glomerular filtration rate (eGFR) calculated by CKD-EPI at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy | Qualitative | 0: No<br>1: Yes |
| Glomerular filtration rate value at week 48 | Value of estimated glomerular filtration rate (eGFR) calculated by CKD-EPI at week 48 (+ or - 2 weeks) of TAF/FTC/BIC therapy | Quantitative, continuous | 1, 1.5, 1.8, 2, n |
| Number of medication claims | Number of TAF/FTC/BIC medication claims during the 48-week follow-up | Quantitative, discrete | 1, 2, 3, n |
| Headache emergency | The patient visited the emergency department during the period of TAF/FTC/BIC use for ICD-10 codes G444 and/or G448 | Qualitative | 0: No<br>1: Yes |
| Diarrhea emergency | The patient visited the emergency department during the period of TAF/FTC/BIC use for ICD-10 code A09X: Diarrhea and gastroenteritis of presumed infectious origin | Qualitative | 0: No<br>1: Yes |
| Nausea and vomiting emergency | The patient visited the emergency department during the period of TAF/FTC/BIC use for ICD-10 code R11X: Nausea and vomiting | Qualitative | 0: No<br>1: Yes |
| Termination of health insurance coverage | The patient terminated their health insurance with EPS SURA. | Qualitative | 0: No<br>1: Yes |
| Date of termination of insurance coverage | Date of termination of health insurance with EPS SURA | Quantitative, continuous | dd/mm/yyyy |
| Death | The patient passed away after the index date | Qualitative | 0: No<br>1: Yes |
| Date of death | Date of patient's death | Quantitative, continuous | dd/mm/yyyy |

## Sample Size

No sampling will be conducted, as data from the entire population (census) that meets the eligibility criteria for this study will be used.

F-INV001 V: 03

## Statistical Analysis

The database created in Access will be transferred to RStudio and Jamovi for the corresponding descriptive analysis.

### Characterization of the Sociodemographic and Clinical Profile

Absolute and relative frequencies will be calculated for categorical variables. For numerical variables, normality will be assessed using the Shapiro-Wilk test. Variables with a p-value greater than 0.05 will be considered to follow a normal distribution and will be represented by means and standard deviations. For variables that do not follow a normal distribution, medians and interquartile ranges will be used.

### **Proportion of Pretreatment Regimens**

The proportion of patients who have received different combinations of ART prior to starting TAF/FTC/BIC will be calculated. Frequency tables will be used to display the proportion of each pretreatment regimen, supplemented by bar charts reflecting the frequencies of the most common treatments.

### Virologic Suppression at 24 and 48 Weeks

Virologic suppression is defined as a viral load of <50 copies/mL at weeks 24 and 48 of treatment. The proportion of patients achieving this threshold will be calculated at both time points, and the results will be compared between weeks 24 and 48 using McNemar's test for related samples.

#### Effective Access to Treatment

Effective treatment is defined as the initiation of therapy within a reasonable time after prescription. The time between prescription and the initiation of treatment will be calculated (mean or median, depending on the normality test), and patients will be classified into two categories: those who initiate treatment effectively (within a short period, generally defined as initiation within 7-14 days of HIV diagnosis) and

F-INV001 V: 03

those who experience delays.

### Paraclinical Results: CD4 T-Lymphocytes, Renal Function, and Lipid Profile

To describe changes in clinical markers at weeks 24 and 48, the summary measure (mean or median, depending on the normality test) of baseline values will be compared with the values of these biomarkers at the two time points. Paired-samples t-tests or Wilcoxon tests will be used if the data distribution is non-normal.

### Rapid Onset of Therapy

The frequency of patients meeting this criterion will be calculated, and the characteristics of those with rapid onset versus those without will be compared using the chi-square test.

### Treatment-Related Adverse Events

Treatment-related adverse events at weeks 24 and 48 will be characterized and classified according to type and severity. The proportion of patients experiencing these events will be calculated and compared between the two time points. Contingency tables and chi-square tests will be used to analyze the relationship between adverse events and other clinical and sociodemographic variables.

## Adherence to Treatment

Adherence will be measured using pharmacy claims information with the Proportion of Days Covered (PDC). PDC calculates the proportion of days the patient has access to the medication over a specified period (64,65). In this study, patients with a PDC of 80% or higher will be considered to have adequate adherence. However, studies have shown that even lower adherence levels can still result in a high rate of viral suppression.

F-INV001 V: 03

### **Biases**

The following biases are considered potential risks in this study:

- Information Bias: This refers to errors introduced during the measurement of exposure, events, and other variables in the study population, which, if present, may lead to erroneous conclusions regarding the hypothesis being investigated. In this study, data obtained from secondary sources such as medical records may not fully or accurately capture the information of interest. To control for this bias, a random review of at least 10% of the clinical histories will be conducted, and the information recorded in the database will be cross-referenced with that found in the clinical records.
- Loss to Follow-up Bias: Loss of participants throughout the study may introduce bias, as the selection of participants is not random.

## Statement on the Application of Ethical Principles in Research

In accordance with Resolution 8430 of 1993, this study is classified as risk-free: it involves retrospective documentary research techniques and methods, with no intervention or intentional modification of the biological, physiological, psychological, or social variables of individuals. The study will be conducted through the review of medical records and will be submitted for approval to the SURA Ethics Committee.

The use of medical records will be in compliance with Resolution 1995 of 1999, ensuring data protection and confidentiality of the information collected. Furthermore, a confidentiality agreement has been signed for academic projects, establishing compliance with legal provisions. This agreement confirms that access to personal data and confidential information from medical records will be provided, data which are considered sensitive under the "habeas data" law. The dissemination of this information could affect the privacy of the data owner. Therefore, all provisions outlined in this document will be strictly adhered to.

F-INV001 V: 03

### **Timeline**

| Activity/Month | 1 | 2 | 3 | 4 | 5 | 6 |
|---------------------|---|---|---|---|---|---|
| Phase 1: | | | | | | |
| Research protocol | | | | | | |
| writing | | | | | | |
| Phase 2: | | | | | | |
| Submission to IRB | | | | | | |
| Phase 3: Execution | | | | | | |
| (analysis and | | | | | | |
| structuring of | | | | | | |
| results and | | | | | | |
| discussion) | | | | | | |
| Phase 4: | | | | | | |
| Technical report | | | | | | |
| writing and closing | | | | | | |
| to IRB | | | | | | |
| Phase 5: Writing of | | | | | | |
| publication-type | | | | | | |
| manuscript and | | | | | | |
| submission to | | | | | | |
| journal and | | | | | | |
| conference | | | | | | |

#### References

- 1. Challacombe SJ. Global inequalities in HIV infection. Oral Dis. 2020 Sep 1;26(S1):16–21.
- 2. del Rio C. The global HIV epidemic: What the pathologist needs to know. Vol. 34, Seminars in Diagnostic Pathology. W.B. Saunders; 2017. p. 314–7.
- 3. Payagala S, Pozniak A. The global burden of HIV. Clin Dermatol. 2024;42(2):119–27.
- 4. Ortblad KF, Lozano R, Murray CJL. The burden of HIV: Insights from the global burden of disease study 2010. Vol. 27, AIDS. 2013. p. 2003–17.
- 5. Fanfair RN, Buchacz K, Peters P. CDC Yellow Book 2024. 2024. Human Immunodeficiency Virus / HIV.
- 6. Bekker LG, Beyrer C, Mgodi N, Lewin SR, Delany-Moretlwe. Sinead, Taiwo B, et al. HIV infection. Nat Rev Dis Primers. 2023;9(1).



- 7. Velasco-Benítez CA. Digestive, Hepatic, and Nutritional Manifestations in Latin American Children With HIV/AIDS. J Pediatr Gastroenterol Nutr. 2008;47:S24–6.
- 8. García PJ, Bayer A, Cárcamo CP. The changing face of HIV in Latin America and the Caribbean. Curr HIV/AIDS Rep. 2014;11(2):146–57.
- 9. Montana JF, Ferreira GRON, Cunha CLF, de Queiroz AAR, Fernandes WAA, Polaro SHI, et al. The HIV epidemic in Colombia: spatial and temporal trends analysis. BMC Public Health. 2021 Dec 1;21(1).
- 10. Rubio-Mendoza ML, Jacobson JO, Morales-Miranda S, Sierra-Alarcón CÁ, Luque-Núñez R. High HIV burden in men who have sex with men across Colombia's largest cities: Findings from an integrated biological and behavioral surveillance study. PLoS One. 2015 Aug 7;10(8).
- 11. Quevedo-Gómez MC, Krumeich A, Abadía-Barrero CE, Van Den Borne HW. Social inequalities, sexual tourism and HIV in Cartagena, Colombia: An ethnographic study. BMC Public Health. 2020 Aug 8;20(1).
- 12. Cuenta de Alto Costo (CAC). Situación del VIH en Colombia, 2023. 2023.
- 13. Toro-Tobón D, Berbesi-Fernández D. Prevalence of HIV/Hepatitis C Virus Co-Infection and Injection Risk Correlations in People Who Inject Drugs in Colombia: A Cross-Sectional Study Using Respondent Driven Sampling. Subst Use Misuse. 2020 Feb 3;55(3):414–23.
- 14. Alzate JC, Pericàs JM, Taylor HA, Benach J. Systemic factors and barriers that hamper adequate data collection on the HIV epidemic and its associated inequalities in countries with long-term armed conflicts: Lessons from Colombia. Am J Public Health. 2018 Oct 1;108(10):1341–4.
- 15. Wirtz AL, Guillén JR, Stevenson M, Ortiz J, Talero MÁB, Page KR, et al. HIV infection and engagement in the care continuum among migrants and refugees from Venezuela in Colombia: a cross-sectional, biobehavioural survey. Lancet HIV. 2023 Jul 1;10(7):e461–71.
- 16. Ministerio de Salud y Protección Social Empresa Nacional Promotora del Desarrollo Territorial ENTerritorio- Instituto de Evaluación Tecnológica en Salud. Guía de Práctica Clínica (GPC) basada en la evidencia científica para la atención de la infección por VIH/SIDA en personas adultas, gestantes y adolescentes. Guía para profesionales de la salud. Guía N° 39-2021. 2021.
- 17. U.S. Department of Health and Human Services Panel on Antiretroviral Guidelines for Adults and Adolescents. Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents With HIV. 2024.
- 18. Markham A. Bictegravir: First Global Approval. Drugs. 2018 Apr 1;78(5):601–6.
- 19. Gutiérrez-Lorenzo M, Rubio-Calvo D, Urda-Romacho J. Effectiveness, safety, and economic impact of the bictegravir/emtricitabine/tenofovir alafenamide regimen in real clinical practice cohort of hiv-1 infected adult patients. Revista Espanola de Quimioterapia. 2021;34(4):315–9.
- Camici M, Gagliardini R, Lanini S, Del Duca G, Mondi A, Ottou S, et al. Rapid ART initiation with bictegravir/emtricitabine/tenofovir alafenamide in individuals presenting with advanced HIV disease (Rainbow study). Int J Antimicrob Agents. 2024 Jan 1;63(1).
- 21. Corona D, Pérez-Valero I, Camacho A, Gutiérrez Liarte Á, Montero-Alonso M, Alemán MR, et al. Effectiveness and safety of bictegravir/emtricitabine/tenofovir alafenamide in HIV late presenters. Int J Antimicrob Agents. 2024 Jan 1;63(1).
- 22. Squillace N, Ricci E, Maggi P, Taramasso L, Menzaghi B, De Socio GV, et al. Real-life safety of Emtricitabine/Tenofovir Alafenamide/Bictegravir. PLoS One. 2023 Aug 1;18(8 August).
- 23. Miller JM, Binnicker MJ, Campbell S, Carroll KC, Chapin KC, Gilligan PH, et al. A Guide to Utilization of the Microbiology Laboratory for Diagnosis of Infectious Diseases: 2018 Update by the Infectious Diseases Society of America and the American Society for Microbiology. Clinical Infectious Diseases. 2018 Aug 31;67(6):e1–94.
- 24. Lucas S, Nelson AM. HIV and the spectrum of human disease. Journal of Pathology. 2015 Jan 1;235(2):229–41.



- 25. Ozorowski G, Pallesen J, De Val N, Lyumkis D, Cottrell CA, Torres JL, et al. Open and closed structures reveal allostery and pliability in the HIV-1 envelope spike. Nature. 2017 Jul 20;547(7663):360–1.
- Chen B. Molecular Mechanism of HIV-1 Entry. Vol. 27, Trends in Microbiology. Elsevier Ltd; 2019.
   p. 878–91.
- 27. Wilen CB, Tilton JC, Doms RW. Molecular mechanisms of HIV entry. Adv Exp Med Biol. 2012;726:223–42.
- 28. Frankel AD, Young JAT. HIV-1: Fifteen Proteins and an RNA [Internet]. Vol. 67, Annu. Rev. Biochem. 2024. Available from: www.annualreviews.org.
- 29. Davenport YW, West AP, Bjorkman PJ. Structure of an HIV-2 gp120 in Complex with CD4. J Virol. 2016 Feb 15;90(4):2112–8.
- 30. Barroso H, Borrego P, Bártolo I, Marcelino JM, Família C, Quintas A, et al. Evolutionary and structural features of the C2, V3 and C3 envelope regions underlying the differences in HIV-1 and HIV-2 biology and infection. PLoS One. 2011;6(1).
- 31. Rosenberg ZF, Fauci AS. Immunopathogenesis of HIV infection [Internet]. Vol. 254, FASEB journal: official publication of the Federation of American Societies for Experimental Biology. 1991. p. 54–64. Available from: www.fasebj.org
- 32. Okoye AA, Picker LJ. CD4+ T-Cell Depletion In Hiv Infection: Mechanisms Of Immunological Failure. Immunol Rev. 2013 Jul;254(1):54–64.
- 33. Vijayan KV, Karthigeyan KP, Tripathi SP, Hanna LE. Pathophysiology of CD4+ T-Cell depletion in HIV-1 and HIV-2 infections. Vol. 8, Frontiers in Immunology. Frontiers Media S.A.; 2017.
- 34. Fauci AS, Pantaleo G, Stanley S, Weissman D. Immunopathogenic Mechanisms of HIV Infection [Internet]. Vol. 124, Ann Intern Med. 1996. Available from: http://annals.org/
- 35. Forsman A, Weiss RA. Why is HIV a pathogen? Trends Microbiol. 2008 Dec;16(12):555–60.
- 36. Moylett EH, Shearer WT. HIV: Clinical manifestations. Vol. 110, Journal of Allergy and Clinical Immunology. Mosby Inc.; 2002. p. 3–16.
- 37. Deeks SG, Overbaugh J, Phillips A, Buchbinder S. HIV infection. Nat Rev Dis Primers. 2015 Oct 1:1.
- 38. Khunnawat C, Mukerji S, Havlichek D, Touma R, Abela GS. Cardiovascular Manifestations in Human Immunodeficiency Virus-Infected Patients. Vol. 102, American Journal of Cardiology. 2008. p. 635–42.
- 39. Ntsekhe M, Baker J V. Cardiovascular Disease among Persons Living with HIV: New Insights into Pathogenesis and Clinical Manifestations in a Global Context. Vol. 147, Circulation. Lippincott Williams and Wilkins; 2023. p. 83–100.
- 40. Vishnu P, Aboulafia DM. Haematological manifestations of human immune deficiency virus infection. Br J Haematol. 2015 Dec 1;171(5):695–709.
- 41. Sereti I, Clifford Lane H. Immunopathogenesis of Human Immunodeficiency Virus: Implications for Immune-Based Therapies. Clin Infect Dis [Internet]. 2001;32(12):1738–55. Available from: http://cid.oxfordjournals.org/
- 42. Guarner J. Human immunodeficiency virus: Diagnostic approach. Vol. 34, Seminars in Diagnostic Pathology. W.B. Saunders; 2017. p. 318–24.
- 43. Walensky RP, Jernigan DB, Bunnell R, Layden J, Kent CK, Gottardy AJ, et al. Sexually Transmitted Infections Treatment Guidelines. Vol. 70, MMWR. Recommendations and reports: Morbidity and mortality weekly report. Recommendations and reports. 2021. p. 1–187.
- 44. Duncan D, Duncan J, Kramer B, Nilsson AY, Haile B, Butcher A, et al. An HIV Diagnostic Testing Algorithm Using the cobas HIV-1/ HIV-2 Qualitative Assay for HIV Type Differentiation and Confirmation. J Clin Microbiol [Internet]. 2021;59(7). Available from: https://www.unaids



- 45. Ministerio de Salud y Protección Social. Guía de Práctica Clínica basada en la evidencia científica para la atención de la infección por VIH/SIDA en personas adultas, gestantes y adolescentes. Guía para profesionales de la salud. Guía Actualización parcial 2021. 2021.
- 46. Cihlar T, Fordyce M. Current status and prospects of HIV treatment. Vol. 18, Current Opinion in Virology. Elsevier B.V.; 2016. p. 50–6.
- 47. Flexner C. Modern Human Immunodeficiency Virus Therapy: Progress and Prospects. Clin Pharmacol Ther. 2019 Jan 1;105(1):61–70.
- 48. Ismail SD, Pankrac J, Ndashimye E, Prodger JL, Abrahams MR, Mann JFS, et al. Addressing an HIV cure in LMIC. Vol. 18, Retrovirology. BioMed Central Ltd; 2021.
- 49. Vella S, Schwartländer B, Sow SP, Eholie SP, Murphy RL. The history of antiretroviral therapy and of its implementation in resource-limited areas of the world. Vol. 26, AIDS. 2012. p. 1231–41.
- 50. Sokhela S, Lalla-Edward S, Siedner MJ, Majam M, Daniel W, Venter F. Roadmap for Achieving Universal Antiretroviral Treatment. Annu Rev Pharmacol Toxicol [Internet]. 2023;63:99–117. Available from: https://sahivsoc.org/Subheader/Index/sahcs-guidelines.
- 51. Alum EU, Uti DE, Ugwu OPC, Alum BN. Toward a cure Advancing HIV/AIDs treatment modalities beyond antiretroviral therapy: A Review. Vol. 103, Medicine (United States). Lippincott Williams and Wilkins; 2024. p. e38768.
- 52. Deeks ED. Bictegravir/emtricitabine/tenofovir alafenamide: A review in HIV-1 infection. Vol. 78, Drugs. Springer International Publishing; 2018. p. 1817–28.
- 53. Tsiang M, Jones GS, Goldsmith J, Mulato A, Hansen D, Kan E, et al. Antiviral activity of bictegravir (GS-9883), a novel potent HIV-1 integrase strand transfer inhibitor with an improved resistance profile. Antimicrob Agents Chemother. 2016 Dec 1;60(12):7086–97.
- 54. Hassounah SA, Alikhani A, Oliveira M, Bharaj S, Ibanescu RI, Osman N, et al. Antiviral Activity of Bictegravir and Cabotegravir against Integrase Inhibitor-Resistant SIVmac239 and HIV-1. Antimicrob Agents Chemother [Internet]. 2017;61(12). Available from: https://doi.org/10.1128/AAC
- 55. Subramanian R, Ling J, Wang J, Wang K, Hao J, Jin H, et al. Human and nonclinical disposition of [14C]bictegravir, a potent integrase strand-transfer inhibitor for the treatment of HIV-1 infection. Xenobiotica. 2022;52(9–11):973–85.
- 56. Gallant J, Lazzarin A, Mills A, Orkin C, Podzamczer D, Tebas P, et al. Bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir, abacavir, and lamivudine for initial treatment of HIV-1 infection (GS-US-380-1489): a double-blind, multicentre, phase 3, randomised controlled non-inferiority trial. The Lancet. 2017 Nov 4;390(10107):2063–72.
- 57. Sax PE, Pozniak A, Montes ML, Koenig E, DeJesus E, Stellbrink HJ, et al. Coformulated bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir with emtricitabine and tenofovir alafenamide, for initial treatment of HIV-1 infection (GS-US-380–1490): a randomised, double-blind, multicentre, phase 3, non-inferiority trial. The Lancet. 2017 Nov 4;390(10107):2073–82.
- 58. De Clercq E, Zhang Z, Huang J, Zhang M, Li G. BikARVTy for the treatment of HIV infection: Progress and prospects. Biochem Pharmacol. 2023;217.
- 59. DailyMed. Label: BIKARVTY- bictegravir sodium, emtricitabine, and tenofovir alafenamide fumarate tablet. 2024.
- 60. Ford N, Migone C, Calmy A, Kerschberger B, Kanters S, Nsanzimana S, et al. Benefits and risks of rapid initiation of antiretroviral therapy. AIDS. 2018 Jan 2;32(1):17–23.
- 61. Dah TTE, Yaya I, Mensah E, Coulibaly A, Kouamé JBM, Traoré I, et al. Rapid antiretroviral therapy initiation and its effect on treatment response in MSM in West Africa. AIDS. 2021 Nov 1;35(13):2201–10.



- 62. Mateo-Urdiales A, Johnson S, Smith R, Nachega JB, Eshun-Wilson I. Rapid initiation of antiretroviral therapy for people living with HIV. Vol. 2019, Cochrane Database of Systematic Reviews. John Wiley and Sons Ltd; 2019.
- 63. Huang YC, Sun HY, Chuang YC, Huang YS, Lin KY, Huang SH, et al. Short-term outcomes of rapid initiation of antiretroviral therapy among HIV-positive patients: Real-world experience from a single-centre retrospective cohort in Taiwan. BMJ Open. 2019 Sep 1;9(9).
- 64. Johns Hopkins Hospital T, Canfield S, Komandt M, Lengel M, Gilmore V, Kilcrease C. Correlation between medication adherence using proportion of days covered and achieving viral suppression in patients living with HIV. Vol. 29, JMCP.org. 2023.
  - 65. de Oliveira Costa J, Zhao Y, Pearson SA, Schaffer AL. Assessing the impact of implementing multiple adherence measures to antiretroviral therapy from dispensing data: a short report. AIDS Care Psychological and Socio-Medical Aspects of AIDS/HIV. 2023;35(7):970–5.